CLINICAL TRIAL: NCT06968052
Title: Effects of Exercise and Feldenkrais Approaches on Position Sense, Strength, Range of Motion and Posture in Cases With Forward Head Posture
Brief Title: Effects of Feldenkrais Approach in Cases With Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC-FTR-Tt25
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Forward Head Posture
Keywords: Rehabilitation; Posture; Proprioception; Exercise; Muscle Strength; Spine
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will employ assessor and statistician blinding. The physiotherapists performing baseline and post-intervention assessments will be blinded to group allocation to minimize bias. Additionally, statistical analyses will be conducted by a researcher blinded to group assignments. Participants and therapists delivering the intervention will not be blinded due to the nature of the exercise-based intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in Group A will receive a combined program of corrective exercises and the Feldenkrais method. The program includes posture-focused Feldenkrais movements and stretching/strengthening exercises for postural muscles (e.g., pectorals, cervical extensors, deep neck flexors, and scapular retractors). The intervention will be delivered twice weekly over 8 weeks, totaling 16supervised 45-minute sessions by a physiotherapist.
  Interventions: Other: Strength and Feldenkrais Exercise
- Group B (Active Comparator): Participants in Group B will receive a program combining corrective and breathing exercises. Corrective exercises will be performed at the same sets and repetitions as Group A, adjusted to individual tolerance. Breathing exercises include diaphragmatic breathing and thoracic expansion, performed in 2-3 sets of 7 repetitions. The intervention will be delivered twice weekly over 8 weeks, totaling 16supervised 45-minute sessions by a physiotherapist.
  Interventions: Other: Strength Exercise

INTERVENTIONS:
Other: Strength and Feldenkrais Exercise — This is a behavioral, non-drug and non-device-based intervention combining somatic awareness through Feldenkrais principles with neuromuscular re-education. Movements emphasize minimal effort, reduced muscle tension, and improved self-perception of posture. The approach supports individualized progression and complements conventional physiotherapy without the use of pharmacological agents or medical equipment.
  Arms: Group A
Other: Strength Exercise — This is a non-drug, non-device corrective exercise program tailored for adults with forward head posture. It includes postural muscle strengthening and stretching, such as deep neck flexor activation, scapular retraction, and pectoral stretching. Additionally, participants perform diaphragmatic and thoracic breathing exercises.
  Arms: Group B

SUMMARY:
It is thought that adding approaches that increase posture awareness to corrective exercise programs will contribute to the treatment. The aim of the study is to evaluate the effect of adding the Feldenkrais method to the corrective exercise program applied to individuals with forward head posture on cervical joint position sense, muscle strength, joint range of motion and posture parameters.

DETAILED DESCRIPTION:
The combination of the Feldenkrais method with corrective exercises stands out as an innovative approach to the problem of forward head posture. This approach aims to not only eliminate physical alignment errors but also increase individuals' internal awareness of posture and movement patterns by integrating traditional postural correction techniques with Feldenkrais' movement efficiency and awareness-oriented principles. In this way, it may be possible for the postural improvements obtained to be more sustainable. It is reported that the Feldenkrais method supports neuromuscular control by increasing body awareness and contributes to movement quality. In light of this information, it is predicted that the addition of the Feldenkrais method to the corrective exercise program applied to individuals with forward head posture will provide additional improvement in cervical joint position sense, muscle strength, range of motion and posture parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age
* CVA (cervicovertebral angle) ≤50° (16,17)
* Spending at least 4 hours of daily desk time 5 days a week

Exclusion Criteria:

* Having temporomandibular dysfunction
* Having any spinal deformity
* Having cervical trauma or pain treatment within the last 6 months
* Having previously participated in a corrective exercise program
* History of neurological disorder
* History of spinal or thoracic surgery
* Having hearing impairment
* Use of analgesics/muscle relaxants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Cervical Joint Position Sense | 8 weeks
  Cervical joint position sense was assessed using a laser pointer-based method to evaluate proprioceptive accuracy. A laser device was securely mounted on the participant's head, and a neutral head position was established as a reference. Participants were instructed to move their heads in specific directions (flexion, extension, lateral flexion, or rotation) and, with eyes closed, return to the starting position. The laser beam projected onto a target screen allowed measurement of repositioning error-the distance between the original and returned laser point. Each direction was tested once, followed by three recorded trials, with the average used for analysis.
Cervical Muscle Strength | 8 weeks
  Cervical muscle strength was assessed isometrically using the Lafayette Manual Muscle Tester. Participants were seated upright in a backless, armless chair with feet flat on the floor. Initial calibration involved maximal voluntary isometric contraction with hands pressed together in front of the body. Measurements were then taken with the neck in a neutral position, applying resistance to the forehead (flexion), occiput (extension), lateral head (lateral flexion), and chin (rotation). Three trials were recorded per direction, with averages used for analysis. A 3-minute rest was provided between attempts. Participants could stop at any time if discomfort occurred.
Cervical Range of Motion | 8 weeks
  Cervical range of motion (ROM) was measured using the Baseline Digital Absolute+Axis Goniometer, a reliable and clinically validated tool for assessing cervical spine movements. Active cervical motions-including flexion, extension, right/left lateral flexion, and right/left rotation-were measured following standardized procedures defined by Norkin et al. Participants performed each movement actively while seated in an upright position. The goniometer provided objective angular measurements. This tool has demonstrated good to excellent intrarater reliability (ICC: 0.70-0.93) in previous research, confirming its suitability for both clinical and research purposes.
Postural Assessment | 8 weeks
  Postural parameters were assessed using the PostureScreen Mobile (PSM) application, a validated digital tool for quantifying postural deviations. Static posture images were taken from anterior, posterior, and lateral views while participants stood in a relaxed upright position. Key anatomical reference points were marked within the app, which then calculated deviations from ideal posture in degrees or centimeters. This method allows for objective and reliable analysis of head, shoulder, and spinal alignment, providing quantifiable data to track changes over time and inform targeted corrective interventions.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 8 weeks
  The Neck Disability Index (NDI) is a self-reported questionnaire designed to evaluate how neck pain affects daily activities. It includes 10 items grouped under pain-related aspects (e.g., pain intensity, headaches, sleep, concentration), selective daily activities (e.g., driving, lifting, work, recreation), and essential daily activities (e.g., personal care, reading). Each item is scored from 0 to 5, and total scores are converted to a percentage out of 100. Higher scores indicate greater disability. The Turkish version of the NDI has demonstrated excellent test-retest reliability (ICC = 0.979) and strong construct validity in Turkish-speaking populations.
Numeric Pain Rating Scale (NPRS) | 8 weeks
  The Numeric Pain Rating Scale (NPRS) is a widely used tool to assess the intensity of pain. Participants are asked to rate their neck pain on a scale from 0 to 10, where 0 indicates "no pain" and 10 represents "the worst pain imaginable." NPRS has demonstrated moderate to high test-retest reliability (ICC = 0.67-0.96) and strong convergent validity (r = 0.79-0.95) when compared with the Visual Analog Scale (VAS). It provides a simple, valid, and reliable measure for both clinical and research purposes in individuals with neck pain.
Global Rating of Change (GROC) Scale | 8 weeks
  The Global Rating of Change (GROC) Scale is a subjective tool used to evaluate participants' perceived change and satisfaction with treatment outcomes. At the end of the intervention period, participants rate their overall change on a 7-point scale ranging from -3 (much worse) to +3 (much better). This measure reflects perceived clinical effectiveness by capturing the individual's overall sense of improvement or deterioration, offering insight into the meaningfulness of treatment from the patient's perspective. The GROC is commonly used in rehabilitation research to complement objective outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa, Istanbul, Buyukcekmece
  - Istanbul University-Cerrahpaşa, Istanbul

IPD SHARING:
Plan to Share IPD: No